CLINICAL TRIAL: NCT06118905
Title: Preserving Geriatric Muscle With an Osteoporosis Medication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY23020192
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Denosumab (Experimental): Denosumab 60mg SQ with placebo zoledronic acid
  Interventions: Drug: Denosumab 60 MG/ML
- Zoledronic acid (Active Comparator): Zoledronic acid 5mg IV with Denosumab placebo
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Infusion

INTERVENTIONS:
Drug: Denosumab 60 MG/ML — Subjects to receive Denosumab 60mg SQ and Zoledronic acid placebo IV
  Other Names: Prolia
  Arms: Denosumab
Drug: Zoledronic Acid 5Mg/Bag 100Ml Infusion — Subjects to receive Zoledronic Acid 5mg IV and Denosumab placebo
  Other Names: Reclast
  Arms: Zoledronic acid

SUMMARY:
Our goal is to demonstrate efficacy of the novel agent Denosumab to improve or preserve muscle health, strength, mobility and function in frail older adults.

DETAILED DESCRIPTION:
Approximately one third of older adults in senior communities fall each year, and falls are the leading cause of morbidity and mortality in this age group. Falls are associated with poor quality of life, disability, and death; the medical cost is over $30 billion annually. Despite these statistics, fall reduction strategies have had limited impact for frail seniors. The most devastating fall-related outcome is a hip or other fracture. Over 90% of hip and nonvertebral fractures occur from a fall, and approximately 85% of long-term care (LTC) residents have osteoporosis. Recently, investigators have reported cross-talk between muscle and bone through mechanical and biochemical pathways. Osteosarcopenia, a newly described geriatric syndrome, involves the coexistence of osteoporosis (low bone mass) and sarcopenia (low muscle mass/function). The coexistence of these conditions puts patients at even greater risk for fall/fracture-related serious adverse outcomes. Denosumab(DEMAB), a medication approved for osteoporosis, acts on molecular targets shared between muscle and bone. In the DEMAB pivotal trial and a meta-analysis in healthy adults, investigators reported a reduction in recalled falls in addition to a decrease in fractures. Therefore, DEMAB has the potential to reduce both falls and fractures in a vulnerable population at high risk for both events. Our goal is to demonstrate efficacy of the novel agent DEMAB to improve or preserve muscle health, strength, mobility and function in frail older adults. If successful, this would lay the groundwork for a larger multicenter trial to examine the dual-action for fall and fracture prevention. To bridge this knowledge gap we propose to conduct a 1-year, randomized, double-blind, active-controlled trial to test the efficacy of DEMAB (expected active muscle agent) versus zoledronic acid (ZOL, muscle control) in at least 155 underserved, LTC, frail institutionalized men and women (age≥65) with osteoporosis. Muscle strength, power, quality, markers, function and bone measures will be collected in a mobile lab. At trial completion, all participants receive ZOL for osteoporosis therapy and to prevent potential bone loss following DEMAB discontinuation. Our objectives include Aim 1: Evaluate efficacy of DEMAB to preserve/improve muscle strength, power, mass and structure. Aim 2: Examine the mechanistic biochemical components of the muscle-bone connection. Aim 3: Explore if the DEMAB effect extends to distal functional outcomes. This study includes a number of innovative features: 1) focus on the neglected LTC population of frail older men and women in whom we have a track record of successful enrollment, 2) inclusion of an approved osteoporosis agent feasible in the LTC setting with a novel focus on muscle strength, power, structure, and function, 3) mobile lab allowing onsite participation, 4) assessment of muscle and bone parameters by portable techniques, and 5) electronic alerts for falls and SAEs. This study will challenge the current paradigm of avoiding anti-fracture/fall therapy in vulnerable fallers and establish the necessary conditions to justify a large trial to maintain muscle and bone health to reduce falls and fractures.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory male and female residents with osteoporosis or low bone mass (at risk for fracture) age 65 and older will be considered if: 1) they reside in an institution (nursing home, assisted living facility or senior community) and; 2) they have osteoporosis as diagnosed by a) BMD (spine, hip or forearm BMD T-score ≤ -2.5 SD), b) a previous adult fragility spine or hip fracture, or c) have osteopenia but would be treated based on FRAX and the BHOF treatment thresholds of a 10-year major fracture risk of ≥ 20% or ≥ 3% hip fracture risk using femoral neck BMD.

Exclusion Criteria:

We will exclude residents with subacute illnesses surviving or those with life expectancy <1 year. We will exclude those currently on a related therapy (including a bisphosphonate, Denosumab, teriparatide, abaloparatide, or romosozumab) or who have been on a bisphosphonate for >1 year during the previous 2 years because some bisphosphonates are long acting. We will exclude subjects with a history of hypocalcemia or contraindication for treatment or those who are on systemic glucocorticoids that may lower muscle strength. We will screen for these conditions by detailed history, chart review, and baseline laboratory analyses. Participants with 25-hydroxyvitamin D levels <25 ng/mL will be treated with vitamin D 50,000 IU/wk for 8 weeks. The patient will be enrolled if the follow-up vitamin D level is 25 ng/mL or more. Patients will be allowed to continue on anticonvulsants because use is common in this population. Women on hormone replacement, raloxifene, or residents prescribed protective hip pads will be allowed to participate and continue on these therapies. We will suggest participants stop calcitonin due to cancer concerns.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Knee extension strength change | 12 Months
  The primary muscle strength outcome measure will be the peak muscle force generated by the dominant leg (same side as dominant hand) knee extensor muscles in the sitting position with the knee at 60 degrees of flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Barnabas Woodlands, Pittsburgh, Pennsylvania, United States